CLINICAL TRIAL: NCT06431035
Title: Effect of Caffeinated Chewing Gum on Dehydration Ability in Bodybuilding Athletes: a Crossover Trial
Brief Title: Caffeine & Bodybuilding Dehydration Ability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chih-Hui Chiu (Other)
Responsible Party: Sponsor-Investigator, Chih-Hui Chiu, Professor, National Taiwan Sport University
Organization: National Taiwan Sport University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 113-3
Record Dates: First submitted 2024-04-08; First posted 2024-05-28 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Caffeine; Placebo
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: The participants were divided into caffeine gum trial (CAF) and placebo trial (PL) with a randomized, double-blind study design.
Who Masked: Investigator
Masking Description: Using placebo chewing gum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caffeine gum (Experimental): Chewing caffeine Gum (CAF trial, containing 5 mg/kg of caffeine) for 10 minutes before test.
  Interventions: Dietary Supplement: caffeine
- placebo (Placebo Comparator): Chewing placebo gum (without caffeine) for 10 minutes before test.
  Interventions: Dietary Supplement: caffeine

INTERVENTIONS:
Dietary Supplement: caffeine — The participants chewed either caffeine gum (5 mg/kg for 10 minutes per chew) or a placebo (10 minutes per chew, using regular gum).
  Other Names: plocabo gum

SUMMARY:
15-20 trained bodybuilding athletes were divided into caffeine gum trial (CAF) and placebo trial (PL) with a randomized, double-blind study design. The participants chewing either caffeine Gum (CAF trial, containing 5 mg/kg of caffeine) or placebo gum (PL) for 10 minutes. After rested for 15 minutes, Participants used the bicycle to adjust the pedal resistance and speed according to their own feelings until they were dehydrated to 2% of their original body weight.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the effect of caffeinated chewing gum on dehydration ability in bodybuilding athletes. Methods: 15-20 trained bodybuilding athletes were divided into caffeine gum trial (CAF) and placebo trial (PL) with a randomized, double-blind study design. The participants chewing either caffeine Gum (CAF trial, containing 5 mg/kg of caffeine) or placebo gum (PL) for 10 minutes. After rested for 15 minutes, Participants used the bicycle to adjust the pedal resistance and speed according to their own feelings until they were dehydrated to 2% of their original body weight. Record time from exercise to completion of dehydration, heart rate, HRV, energy expenditure, fat oxidation rate and carbohydrate oxidation rate.

ELIGIBILITY:
Inclusion Criteria:

* having won the top 8 places in a national competition,
* having no cardiovascular or joint diseases
* being an adult male

Exclusion Criteria:

* no top 8 finishes at national level
* cardiovascular or joint disease, or any other condition that could be impaired by exercise
* female and underage participants
* previous caffeine allergy

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
dehydration speed | 15 minutes after intervention
  The participants start dehydration until dehydrated to 2% of their original body weight.

SECONDARY OUTCOMES:
energy expenditure | 15 minutes after intervention
  The energy expenditure during dehydration

CONTACTS AND LOCATIONS:
Overall Officials: ChihHui Chiu, PhD, Principal Investigator — National Taiwan University of Sport
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Only participant number and experimental data are provided.

REFERENCES:
- [Derived] Liu HS, Okada T, Mitsuya H, Hsieh MH, Hou CW, Chang CC, Chiu CH. Effects of caffeinated chewing gum-induced sympathetic activation and diuretic effect on the rapid rate of weight loss in bodybuilders: a double-blind crossover study. BMC Sports Sci Med Rehabil. 2025 Apr 26;17(1):98. doi: 10.1186/s13102-025-01144-z. PMID 40287780

DOCUMENTS (1):
  • Study Protocol (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT06431035/Prot_000.pdf